CLINICAL TRIAL: NCT02786901
Title: A Phase 3, Multi-Center, Double-Masked, Vehicle-Controlled, Randomized, Parallel-Group Study to Assess Loteprednol Etabonate Ophthalmic Gel, (BID and TID) Versus Vehicle Gel
Brief Title: LE Gel for the Treatment of Ocular Inflammation and Pain Following Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 875
Record Dates: First submitted 2016-05-23; First posted 2016-06-01 (Estimated); Results first posted 2020-04-14 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Cataract; Pain; Ocular Inflammation
MeSH Terms: conditions — Cataract; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Loteprednol Etabonate Ophthalmic Gel dosed TID (Experimental): Gel
  Interventions: Drug: Loteprednol Etabonate Ophthalmic Gel dosed TID
- Loteprednol Etabonate Ophthalmic Gel dosed BID (Experimental): Gel
  Interventions: Drug: Loteprednol Etabonate Ophthalmic Gel dosed BID
- Vehicle Gel (Placebo Comparator): Vehicle
  Interventions: Drug: Vehicle Gel

INTERVENTIONS:
Drug: Loteprednol Etabonate Ophthalmic Gel dosed TID — Gel
  Other Names: LE
  Arms: Loteprednol Etabonate Ophthalmic Gel dosed TID
Drug: Loteprednol Etabonate Ophthalmic Gel dosed BID — Gel
  Other Names: LE
  Arms: Loteprednol Etabonate Ophthalmic Gel dosed BID
Drug: Vehicle Gel — Gel
  Other Names: Vehicle
  Arms: Vehicle Gel

SUMMARY:
Loteprednol Etabonate Ophthalmic Gel, (BID and TID) versus Vehicle Group for the Treatment of Ocular Inflammation and Pain Following Cataract Surgery.

DETAILED DESCRIPTION:
A Phase 3, Multi-Center, Double-Masked, Vehicle Controlled, Randomized, Parallel-Group Study to Assess Loteprednol Etabonate Ophthalmic Gel, (BID and TID) versus Vehicle Group for the Treatment of Ocular Inflammation and Pain Following Cataract Surgery.

ELIGIBILITY:
Key Inclusion Criteria:

1. Be 18 years or older on the date the Informed Consent Form (ICF) is signed and with the capacity to provide voluntary informed consent.
2. Be able to read, understand, and provide written informed consent on the Institutional Review Board (IRB)/Ethics Committee (EC) approved ICF and provide Health Insurance Portability and Accountability Act (HIPAA) authorization.
3. Be willing and able to comply with all treatment and follow-up/study procedures.
4. Be a candidate for routine, uncomplicated cataract surgery (phaco-emulsification with posterior chamber intraocular lens [IOL] implantation, not combined with any other surgery).
5. In the Investigator's opinion, have potential postoperative pin-holed Snellen visual acuity (VA) of at least 20/200 in the study eye at Visit 1 (Screening) and at least 20/200 in the fellow eye.

Key Exclusion Criteria:

1. Have a severe/serious ocular condition or history/presence of chronic generalized systemic disease that the Investigator feels might increase the risk to the subject or confound the result(s) of the study.
2. Be a female subject who is pregnant or breastfeeding.
3. Be monocular (fellow eye is nonfunctional or fellow eye's pinhole vision is worse than Snellen 20/200).
4. Have had ocular surgery (including laser surgery) in the study eye within 3 months or in the fellow eye within 2 weeks prior to Visit 1 (Screening).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-06-13 (Actual); Study Completion 2017-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise Ramjit, Study Director — Valeant Pharmaceuticals
Locations (6):
- United States (6):
  - Valeant Site 01, Phoenix, Arizona
  - Valeant Site 03, Oceanside, California
  - Valeant Site 05, Miami, Florida
  - Valeant Site 04, Quincy, Massachusetts
  - Valeant Site 06, Kansas City, Missouri
  - Valeant Site 02, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Vehicle BID and TID: Vehicle Gel dosed BID and Vehicle Gel dosed TID, combined
- LE Gel BID: Loteprednol Etabonate Ophthalmic Gel dosed BID
- LE Gel TID: Loteprednol Etabonate Ophthalmic Gel dosed TID
Period: Overall Study
Arm/Group | Vehicle BID and TID | LE Gel BID | LE Gel TID
Started | 199 | 201 | 200
Completed | 122 | 145 | 159
Not Completed | 77 | 56 | 41
Not completed — Adverse Event | 1 | 1 | 2
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Rescue Therapy Use | 71 | 49 | 33
Not completed — Subject Request/Lost to Follow up | 1 | 5 | 5
Not completed — Disallowed medication | 1 | 1 | 0
Not completed — Randomized in error | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle BID and TID | LE Gel BID | LE Gel TID | Total
Number analyzed (Participants) | 199 | 201 | 200 | 600
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (8.92) | 68.3 (9.11) | 67.9 (9.32) | 68.2 (9.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 117 | 130 | 363
  Male | 83 | 84 | 70 | 237
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 7 | 13 | 9 | 29
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 14 | 23 | 23 | 60
  White | 169 | 158 | 163 | 490
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 9 | 4 | 3 | 16
Iris Color [Count of Participants; unit: Participants]
  Blue | 50 | 47 | 49 | 146
  Brown | 111 | 115 | 112 | 338
  Green | 17 | 9 | 5 | 31
  Hazel | 20 | 28 | 32 | 80
  Other | 1 | 2 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Resolution of Anterior Chamber (AC) Cells at Visit 5 (Postoperative Day 8)
Description: Slit lamp examination was performed. White blood cell accumulation in anterior aqueous humor was assessed by the Investigator during slit lamp examination and graded on a 5-point scale: Grade 0 = no cells seen; Grade 1 = 1 to 5 cells; Grade 2 = 6 to 15 cells; Grade 3 = 16 to 30 cells; Grade 4 = > 30 cells. Complete resolution of AC cells was defined as Cell score = 0 in the study eye.
Time Frame: 8 days
Population: Missing values and post rescue values imputed as failures.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle BID and TID | LE Gel BID | LE Gel TID
Number analyzed (Participants) | 199 | 201 | 200
Participants | 40 | 52 | 61

2. Primary Outcome: Number of Participants With Complete Resolution of Ocular Pain in Study Eye at Visit 5 (Postoperative Day 8)
Description: Ocular pain, defined as a positive sensation of the eye, including foreign body sensation, stabbing, throbbing, or aching, was assessed and graded by subjects on a 6-point scale: 0 (None), 1 (Minimal), 2 (Mild), 3 (Moderate), 4 (Moderately Severe), and 5 (Severe). Complete Resolution of Ocular Pain was defined as Pain Score = 0.
Time Frame: 8 days
Population: Missing values and post rescue values imputed as failures.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle BID and TID | LE Gel BID | LE Gel TID
Number analyzed (Participants) | 199 | 201 | 200
Participants | 99 | 151 | 151

3. Secondary Outcome: Number of Participants With Complete Resolution of Anterior Chamber (AC) Cells in the Study Eye at Final On-treatment Visit.
Description: as for outcome 1
Time Frame: 14 days
Population: Missing values and post rescue values imputed as failures.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle BID and TID | LE Gel BID | LE Gel TID
Number analyzed (Participants) | 190 | 201 | 198
Participants | 67 | 82 | 94

4. Secondary Outcome: Number of Participants With Complete Resolution of Ocular Pain in Study Eye at Final On-Treatment Visit
Description: as for outcome 2
Time Frame: 14 days
Population: Missing values and post rescue values imputed as failures.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle BID and TID | LE Gel BID | LE Gel TID
Number analyzed (Participants) | 190 | 201 | 198
Participants | 122 | 168 | 170

5. Secondary Outcome: Number of Participants With Complete Resolution of Anterior Chamber (AC) Flare in the Study Eye at Final On-Treatment Visit
Description: Flare was evaluated by the Investigator by assessing the scattering of a slit lamp light beam directed into the anterior chamber (Tyndall effect). Flare was graded on a 5-point scale: 0 (None), 1 (Mild), 2 (Moderate), 3 (Severe), and 4 (Very Severe). An AC flare score of 0 in the study eye was considered complete resolution.
Time Frame: 14 days
Population: Missing values and post rescue values imputed as failures.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle BID and TID | LE Gel BID | LE Gel TID
Number analyzed (Participants) | 190 | 201 | 198
Participants | 107 | 143 | 153

6. Secondary Outcome: Number of Participants With Complete Resolution of Both Anterior Chamber (AC) Cells and AC Flare in the Study Eye at Final On-Treatment Visit
Description: Slit lamp examination was performed. White blood cell accumulation in anterior aqueous humor was assessed by the Investigator during slit lamp examination and graded on a 5-point scale: Grade 0 = no cells seen; Grade 1 = 1 to 5 cells; Grade 2 = 6 to 15 cells; Grade 3 = 16 to 30 cells; Grade 4 = > 30 cells. Complete resolution of AC cells was defined as Cell score = 0 in the study eye. Flare was evaluated by the Investigator by assessing the scattering of a slit lamp light beam directed into the anterior chamber (Tyndall effect). Flare was graded on a 5-point scale: 0 (None), 1 (Mild), 2 (Moderate), 3 (Severe), and 4 (Very Severe). An AC flare score of 0 in the study eye was considered complete resolution.
Time Frame: 14 days
Population: Missing values and post rescue values imputed as failures.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle BID and TID | LE Gel BID | LE Gel TID
Number analyzed (Participants) | 190 | 201 | 198
Participants | 66 | 82 | 92

7. Secondary Outcome: Change From Baseline in Summed Anterior Chamber (AC) Cell and Flare Scores at Final On-Treatment Visit
Description: Slit lamp examination was performed. White blood cell accumulation in anterior aqueous humor was assessed by the Investigator during slit lamp examination and graded on a 5-point scale: Grade 0 = no cells seen; Grade 1 = 1 to 5 cells; Grade 2 = 6 to 15 cells; Grade 3 = 16 to 30 cells; Grade 4 = > 30 cells. Flare was evaluated by the Investigator by assessing the scattering of a slit lamp light beam directed into the anterior chamber (Tyndall effect). Flare was graded on a 5-point scale: 0 (None), 1 (Mild), 2 (Moderate), 3 (Severe), and 4 (Very Severe). The combined endpoint was defined as the sum of the scores for AC cells and AC flare. Summed Anterior Chamber (AC) Cell and Flare Scores could range from 0 to 8.
Time Frame: 14 days
Population: Missing values and post-rescue values imputed using last observation carried forward.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vehicle BID and TID | LE Gel BID | LE Gel TID
Number analyzed (Participants) | 190 | 201 | 198
score on a scale | -1.2 (1.90) | -2.0 (1.50) | -2.1 (1.50)

8. Secondary Outcome: Number of Participants With Treatment Failure at Visit 5 (Postoperative Day 8)
Description: A participant was considered a treatment failure at Visit 5 if they started any rescue medication prior to, or on the day of, Visit 5. If a subject did not have a Visit 5, due either to early discontinuation or to a missed visit, then treatment failure at Visit 5 was defined as starting rescue medication prior to, or on, Postoperative Day 8.
Time Frame: 8 days
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle BID and TID | LE Gel BID | LE Gel TID
Number analyzed (Participants) | 199 | 201 | 200
Participants | 62 | 23 | 20

ADVERSE EVENTS:
Time Frame: 14 days
Description: The Safety population was used for reporting of adverse events. One participant was included in the vehicle group in the ITT (Intent to Treat) population but did not administer study drug, so this participant was excluded from the Safety population. Another participant, randomized to the LE gel TID group, and included in this treatment group in the ITT population, actually received LE gel BID and so was included in LE gel BID treatment group in the Safety population
Arm/Group | Vehicle BID and TID | LE Gel BID | LE Gel TID
All-Cause Mortality (participants affected / at risk) | 0/198 | 0/202 | 0/199
Serious Adverse Events (participants affected / at risk) | 1/198 | 0/202 | 0/199
Other Adverse Events (participants affected / at risk) | 0/198 | 0/202 | 0/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle BID and TID (N=198) | LE Gel BID (N=202) | LE Gel TID (N=199)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor directly for additional information.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT02786901/Prot_SAP_000.pdf